CLINICAL TRIAL: NCT00893126
Title: Premature Coronary Artery Disease (CAD) in Severe Psoriasis
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Prachi P Agarwal, M.D., Principal Investigator, University of Michigan
Other Study IDs: HUM00020514
Record Dates: First submitted 2009-05-01; First posted 2009-05-05 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Psoriasis; Coronary Artery Disease
Keywords: psoriasis; coronary arteriosclerosis; coronary events; rheumatoid arthritis; arthritis
MeSH Terms: conditions — Psoriasis; Coronary Artery Disease; Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 31 ml of blood will be drawn in conjunction with this study.Lipid, Glucose and Lipoprotein will be drawn in one SST tube = 7 ml. Insulin (INS) will be collected in one Green top tube = 7 ml. HSCRP- will be collected in on SSS tube = 7 ml. IL-6 will be collected in Red or Lavender top tube = 7 ml. An additional 3 ml will be drawn for ICAM testing. (The blood for the ICAM testing and IL- 6 will be drawn and frozen until funding has been obtained to run these tests). Specimens will be be properly disposed of after testing is completed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects with severe psoriasis: Subjects 18 to 55 with severe psoriasis. Subject will undergo a CCTA (Coronary CT Angiogram) scan.
  Interventions: Procedure: CCTA Scan (Coronary CT Angiogram)
- Subjects without psoriasis: Subjects 18 to 55 who do not have psoriasis or rheumatologic conditions, including rheumatoid arthritis and systemic lupus erythematosus. This group of subjects will complete a CCTA (Coronary CT Angiogram)scan.
  Interventions: Procedure: CCTA Scan (Coronary CT Angiogram)

INTERVENTIONS:
Procedure: CCTA Scan (Coronary CT Angiogram) — CCTA scan will be performed to study and evaluate the prevalence and severity of coronary artery disease (CAD).

SUMMARY:
The purpose of this study is to compare the prevalence and severity of CAD (coronary artery disease) in patients with and without severe psoriasis, otherwise matched for cardiovascular risk factors.

DETAILED DESCRIPTION:
To establish the relationship between psoriasis and coronary disease by comparing the prevalence and severity of CAD (coronary artery disease) in patients with and without severe psoriasis, otherwise matched for cardiovascular risk factors, as determined by CT coronary calcium scoring and Coronary CT angiography.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe psoriasis as determined by more than two episodes of systemic or inpatient treatment and 10% or more body surface area involvement.
2. Male or female ages 18 to 55 (because CAD risk has been shown to be greatest in younger psoriasis patients in earlier studies, this pilot study will focus on young individuals).
3. Able to give informed consent

Exclusion Criteria:

1. Prior diagnosis of CAD (coronary artery disease) or heart disease based upon one or more of the following:

   * coronary arteriography
   * percutaneous coronary intervention
   * cardiac surgery including bypass graft surgery
   * valve surgery
   * congenital heart disease repair
   * stress ECG or imaging
   * myocardial infarction
   * angina or unstable angina
   * congestive heart failure
   * cardiomyopathy
2. History of anti-oxidants such as fish oil or biologic therapy Tumor Necrosis Factor alpha inhibitors (such as etanercept, adalimumab, or infliximab). A recent review by Sattar et al [22] has shown preliminary evidence that TNF (tumor necrosis factor) blockade can modulate nontraditional cardiovascular risk factors such as C-reactive protein(CRP), Interleukin-6(IL-6), Apolipoprotein AI(ApoAI), Lipoprotein(a)(Lp[a]), Sex Hormone Binding Globulin (SHBG), and homocysteine to exert a possible vascular and metabolic protective effect.
3. Pustular and erythrogenic psoriasis
4. Unable to give informed consent
5. Contraindications to coronary CT, including:

   * Irregular heart rate, such as multiple PVCs (premature ventricular contractions), atrial fibrillation
   * Active heart failure
   * Serum creatinine > 1.5mg/dl
   * Weight > 320 lbs (due to degradation in CT (computerized tomography)image quality by image noise)
   * History of severe allergy to intravenous contrast media
   * High irregular heart rate with contraindications to beta-blockers
   * Pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects with severe psoriasis will be selected prospectively from the clinics of the University of Michigan, Dept. of Dermatology.
  The comparison group (subjects without psoriasis) will be targeted in the Dermatology clinic by screening for matching variables before enrollment. This group will be matched by age and gender to the psoriasis population, and on Framingham risk score.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2009-11; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
To establish the relationship between psoriasis and coronary disease | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Prachi P Agarwal, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No